CLINICAL TRIAL: NCT05104281
Title: Osimertinib Combined With Bevacizumab in Patients With Brain Metastasis Epidermal Growth Factor Receptor (EGFR) Mutation Positive Metastatic Non-Small Cell Lung Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qingdao Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QDCH2021-10-01
Record Dates: First submitted 2021-10-21; First posted 2021-11-02 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Bronchial Neoplasms; EGFR Mutation; Osimertinib; Bevacizumab
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Bronchial Neoplasms | interventions — osimertinib; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- study drug (Experimental): osimertinib 80 mg, oral daily and bevacizumab 15mg/KG body weight intravenously infusion every 21 days
  Interventions: Drug: osimertinib oral and bevazizumab intravenously

INTERVENTIONS:
Drug: osimertinib oral and bevazizumab intravenously — osimertinib 80mg, oral daily and bevacizumab 15mg/KG body weight intravenously infusion every 21 days.
  Other Names: bevacizumab; osimertinib

SUMMARY:
There is no positive data on osimertinib in the treatment of metastatic EGFR mutation positive non-small-cell lung cancer (NSCLC). The purpose of this study is to study osimertinib combined with bevacizumab in the management of patients with brain metastasis harboring EGFR mutation.

DETAILED DESCRIPTION:
Lung cancer is one of the most common types of cancer and is the most common cause of death from cancer (almost 20 percent [%] of cancer deaths); NSCLC accounts for 80% to 85% of lung cancers. The hypothesis is that osimertinib combined bevacizumab in patients with advanced NSCLC patients with brain metastasis characterized by EGFR mutations . Efficacy assessments will include disease assessment, symptomatic progression and patient-reported outcome. Safety assessments will include physical examinations, vital signs, electrocardiograms (ECGs), Eastern Cooperative Oncology Group (ECOG) performance status and clinical safety laboratory assessments (serum chemistry, hematology, coagulation, and urinalysis).

ELIGIBILITY:
Inclusion Criteria:

Participant must have histologically or cytologically confirmed, metastatic, nonsquamous non-small cell lung cancer (NSCLC) Partipiant harboring primary epidermal growth factor receptor (EGFR) Exon 18-21 mutation and brain metastasis.

Participant must have measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.

Participant must have Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1, or 2.

Participant must agree to genetic characterization of tumor status through the required pretreatment tumor biopsy (or submission of equivalent archival material), as well as baseline and periodic blood samples for analysis of tumor mutations in the bloodstream.

A female participant of childbearing potential must have a negative serum or urine test at screening and within 72 hours of the first dose of study treatment and must agree to further serum or urine pregnancy tests during the study.

Exclusion Criteria:

Participant has history of spinal cord compression that has not been treated definitively with surgery or radiation.

Participant has a medical history of interstitial lung disease (ILD), including drug-induced ILD, or radiation pneumonitis.

Participant has a contraindication to the use Osimertinib or Bevacizumab.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS | 30 months
  Progression-Free Survival (PFS) According to RECIST v1.1 as Assessed by Blinded Independent Central Review (BICR)

SECONDARY OUTCOMES:
OS | Up to 48 months
  Overall Survival is defined as the time from the date of randomization to the date of participant's death due to any cause.
ORR | Up to 48 months
  ORR is defined as the percentage of participants who achieve either a complete response (CR) or partial response (PR) as defined by BICR using RECIST v1.1 criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Qingdao Central Hospital, Qingdao Cancer Hospital, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Zhang L, You Y, Liu X, Liu F, Nie K, Ji Y. Osimertinib combined with bevacizumab as the first-line treatment in non-small cell lung cancer patients with brain metastasis harboring epidermal growth factor receptor mutations. Thorac Cancer. 2023 May;14(15):1355-1361. doi: 10.1111/1759-7714.14880. Epub 2023 Apr 5. PMID 37016906